CLINICAL TRIAL: NCT01012739
Title: A Randomized, Partially-blinded, Single-dose, 4-way Cross-over Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Orally Inhaled Indacaterol Maleate Administered Via the Concept1 Device or Via the Simoon Device
Brief Title: Efficacy, Safety, Tolerability, and Pharmacokinetics of Indacaterol Maleate Via Concept1 or Simoon Devices
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQAB149B2222; 2009-012600-48 (EudraCT Number)
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Asthma
Keywords: asthma; QAB149; indacaterol; pulmonary function
MeSH Terms: conditions — Asthma | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Indacaterol 150μg-placebo-Indacaterol 60μg-Indacaterol 120μg (Experimental): In treatment period 1, patients received indacaterol 150 μg via the Concept1 dry-powder inhaler (DPI); in treatment period 2, patients received placebo to indacaterol via the Concept1 DPI; in treatment period 3, patients received indacaterol 60 μg via the Simoon DPI; and in treatment period 4, patients received indacaterol 120 μg via the Simoon DPI. Patients received each treatment only once. There was a washout period of 14-17 days between treatments for patients undergoing pharmacokinetic (PK) assessments; for patients not undergoing PK assessments, the washout period was 7-10 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg via the Concept1 dry-powder inhaler; Drug: Indacaterol 60 μg via the Simoon dry-powder inhaler; Drug: Indacaterol 120 μg via the Simoon dry-powder inhaler; Drug: Placebo to indacaterol via the Concept1 dry-powder inhaler
- Indacaterol 60μg-Indacaterol 150μg-Indacaterol 120μg-placebo (Experimental): In treatment period 1, patients received indacaterol 60 μg via the Simoon dry-powder inhaler (DPI); in treatment period 2, patients received indacaterol 150 μg via the Concept1 DPI; in treatment period 3, patients received indacaterol 120 μg via the Simoon DPI; and in treatment period 4, patients received placebo to indacaterol via the Concept1 DPI. Patients received each treatment only once. There was a washout period of 14-17 days between treatments for patients undergoing pharmacokinetic (PK) assessments; for patients not undergoing PK assessments, the washout period was 7-10 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg via the Concept1 dry-powder inhaler; Drug: Indacaterol 60 μg via the Simoon dry-powder inhaler; Drug: Indacaterol 120 μg via the Simoon dry-powder inhaler; Drug: Placebo to indacaterol via the Concept1 dry-powder inhaler
- Indacaterol 120μg-Indacaterol 60μg-placebo-Indacaterol 150μg (Experimental): In treatment period 1, patients received indacaterol 120 μg via the Simoon dry-powder inhaler (DPI); in treatment period 2, patients received indacaterol 60 μg via the Simoon DPI; in treatment period 3, patients received placebo to indacaterol via the Concept1 DPI; and in treatment period 4, patients received indacaterol 150 μg via the Concept1 DPI. Patients received each treatment only once. There was a washout period of 14-17 days between treatments for patients undergoing pharmacokinetic (PK) assessments; for patients not undergoing PK assessments, the washout period was 7-10 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg via the Concept1 dry-powder inhaler; Drug: Indacaterol 60 μg via the Simoon dry-powder inhaler; Drug: Indacaterol 120 μg via the Simoon dry-powder inhaler; Drug: Placebo to indacaterol via the Concept1 dry-powder inhaler
- Placebo-Indacaterol 120μg- Indacaterol 150μg- Indacaterol 60μg (Experimental): In treatment period 1, patients received placebo to indacaterol via the Concept1 dry-powder inhaler (DPI); in treatment period 2, patients received indacaterol 120 μg via the Simoon DPI; in treatment period 3, patients received indacaterol 150 μg via the Concept1 DPI; and in treatment period 4, patients received indacaterol 60 μg via the Simoon DPI. Patients received each treatment only once. There was a washout period of 14-17 days between treatments for patients undergoing pharmacokinetic (PK) assessments; for patients not undergoing PK assessments, the washout period was 7-10 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg via the Concept1 dry-powder inhaler; Drug: Indacaterol 60 μg via the Simoon dry-powder inhaler; Drug: Indacaterol 120 μg via the Simoon dry-powder inhaler; Drug: Placebo to indacaterol via the Concept1 dry-powder inhaler

INTERVENTIONS:
Drug: Indacaterol 150 μg via the Concept1 dry-powder inhaler — Indacaterol maleate 150 μg was provided in powder filled capsules with the Concept1 dry-powder inhaler.
Drug: Indacaterol 60 μg via the Simoon dry-powder inhaler — Indacaterol 60 μg was provided in powder filled capsules with the Simoon dry-powder inhaler.
Drug: Indacaterol 120 μg via the Simoon dry-powder inhaler — Indacaterol 120 μg was provided in powder filled capsules with the Simoon dry-powder inhaler.
Drug: Placebo to indacaterol via the Concept1 dry-powder inhaler — Placebo to indacaterol was provided in powder filled capsules with the Concept1 dry-powder inhaler.

SUMMARY:
This study assessed the efficacy, safety, tolerability, and pharmacokinetics of two different formulations of indacaterol, one administered via the Concept1 device and one administered via the Simoon device. The study aimed to determine whether the novel formulation (Simoon) had a similar profile to that of the established formulation (Concept1).

DETAILED DESCRIPTION:
This study was double-blind with regards to the Concept1, where placebo for the lactose-blended indacaterol was available. However, with regards to the Simoon, neither the subject nor the investigator was blinded due to lack of a placebo to the PulmoSphere formulation. Hence, the overall designation of the study was partially-blind.

ELIGIBILITY:
Inclusion criteria:

* Patients with persistent asthma with a forced expiratory volume in 1 second (FEV1) ≥ 50%
* Patients using inhaled corticosteroid (with or without long-acting beta agonist)

Exclusion criteria:

* Asthma exacerbations in previous 6 months
* Chronic obstructive pulmonary disease (COPD) or other pulmonary disease
* Excessive use of short-acting beta agonists

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Groningen, Netherlands
- United Kingdom (2):
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Manchester

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Indacaterol 150μg-placebo-Indacaterol 60μg-Indacaterol 120μg | Indacaterol 60μg-Indacaterol 150μg-Indacaterol 120μg-placebo | Indacaterol 120μg-Indacaterol 60μg-placebo-Indacaterol 150μg | Placebo-Indacaterol 120μg- Indacaterol 150μg- Indacaterol 60μg
Started | 9 | 8 | 9 | 9
Completed | 9 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Treatment Period 2
Arm/Group | Indacaterol 150μg-placebo-Indacaterol 60μg-Indacaterol 120μg | Indacaterol 60μg-Indacaterol 150μg-Indacaterol 120μg-placebo | Indacaterol 120μg-Indacaterol 60μg-placebo-Indacaterol 150μg | Placebo-Indacaterol 120μg- Indacaterol 150μg- Indacaterol 60μg
Started | 9 | 8 | 9 | 8
Completed | 9 | 8 | 9 | 7
Not Completed | 0 | 0 | 0 | 1
Not completed — Abnormal test procedure results | 0 | 0 | 0 | 1
Period: Treatment Period 3
Arm/Group | Indacaterol 150μg-placebo-Indacaterol 60μg-Indacaterol 120μg | Indacaterol 60μg-Indacaterol 150μg-Indacaterol 120μg-placebo | Indacaterol 120μg-Indacaterol 60μg-placebo-Indacaterol 150μg | Placebo-Indacaterol 120μg- Indacaterol 150μg- Indacaterol 60μg
Started | 9 | 8 | 9 | 7
Completed | 9 | 8 | 9 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Indacaterol 150μg-placebo-Indacaterol 60μg-Indacaterol 120μg | Indacaterol 60μg-Indacaterol 150μg-Indacaterol 120μg-placebo | Indacaterol 120μg-Indacaterol 60μg-placebo-Indacaterol 150μg | Placebo-Indacaterol 120μg- Indacaterol 150μg- Indacaterol 60μg
Started | 9 | 8 | 9 | 7
Completed | 9 | 8 | 9 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: The entire study population included all 4 treatment groups who received indacaterol 150 µg via the Concept1 dry-powder inhaler (DPI), indacaterol 60 µg via the Simoon DPI, indacaterol 120 µg via the Simoon DPI, and placebo to indacaterol via the Concept1 DPI. Patients received each treatment only once. There was a washout period of 14-17 days between treatments for patients undergoing pharmacokinetic (PK) assessments; for patients not undergoing PK assessments, the washout period was 7-10 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 35
Age Continuous [Mean (Standard Deviation); unit: years] | 42.6 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose for Each Treatment
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose for each treatment.
Time Frame: Baseline and Day 1
Population: Pharmacodynamic analysis set: All randomized patients that received at least 1 dose of study drug and had a baseline and at least 1 post-baseline measurement of FEV1.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Indacaterol 150 μg: Patients received indacaterol 150 μg via the Concept1 dry-powder inhaler (DPI) only once. There was a washout period of 14-17 days between treatments for patients undergoing pharmacokinetic (PK) assessments; for patients not undergoing PK assessments, the washout period was 7-10 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
- Indacaterol 60 μg: Patients received Indacaterol 60 μg via the Simoon dry-powder inhaler only once. There was a washout period of 14-17 days between treatments for patients undergoing pharmacokinetic (PK) assessments; for patients not undergoing PK assessments, the washout period was 7-10 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
- Indacaterol 120 μg: Patients received Indacaterol 120 μg via the Simoon dry-powder inhaler only once. There was a washout period of 14-17 days between treatments for patients undergoing pharmacokinetic (PK) assessments; for patients not undergoing PK assessments, the washout period was 7-10 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
- Placebo to Indacaterol: Patients received placebo to indacaterol via the Concept1 dry-powder inhaler only once. There was a washout period of 14-17 days between treatments for patients undergoing pharmacokinetic (PK) assessments; for patients not undergoing PK assessments, the washout period was 7-10 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
Arm/Group | Indacaterol 150 μg | Indacaterol 60 μg | Indacaterol 120 μg | Placebo to Indacaterol
Number analyzed (Participants) | 33 | 33 | 34 | 35
Liters | 2.97 (0.695) | 2.93 (0.688) | 2.91 (0.734) | 2.77 (0.67)

2. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (FEV1) for Each Treatment
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5, 15, and 30 minutes; and 1, 2, 4, 6, 8, and 12 hours post-dose in Day 1.
Time Frame: Baseline and Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Indacaterol 150 μg | Indacaterol 60 μg | Indacaterol 120 μg | Placebo to Indacaterol
Number analyzed (Participants) | 33 | 33 | 34 | 35
Liters | 3.19 (0.747) | 3.15 (0.745) | 3.15 (0.717) | 2.96 (0.682)

3. Secondary Outcome: Time to Peak Forced Expiratory Volume in 1 Second (FEV1) for Each Treatment
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards at 5, 15, and 30 minutes; 1 hour, 1 hour 30 minutes; and 1, 2, 4, 6, 8, and 12 hours post-dose in Day 1.
Time Frame: From 5 minutes to 12 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Indacaterol 150 μg | Indacaterol 60 μg | Indacaterol 120 μg | Placebo to Indacaterol
Number analyzed (Participants) | 33 | 33 | 34 | 35
Hours | 6.80 (7.614) | 8.22 (7.990) | 7.50 (7.370) | 7.93 (7.747)

4. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 4 Hours Post-dose for Each Treatment
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5, 15, and 30 minutes; and 1, 2, and 4 hours post-dose. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time.
Time Frame: From 5 minutes to 4 hours post-dose for each treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Indacaterol 150 μg | Indacaterol 60 μg | Indacaterol 120 μg | Placebo to Indacaterol
Number analyzed (Participants) | 33 | 33 | 34 | 35
Liters | 3.03 (0.743) | 2.96 (0.732) | 2.99 (0.722) | 2.78 (0.651)

5. Secondary Outcome: Indacaterol Exposure (AUC[0-24 Hours]) for Each Treatment
Description: All patients fasted for at least 10 hours prior to administration of study medication and continued to fast for at least 4 hours thereafter. Venous blood samples for pharmacokinetic evaluation were collected at 5, 10, 15, and 30 minutes; and 1, 2, 4, 8, and 24 hours post-dose in each treatment period and were analyzed using a LC-MS/MS assay. Area under the concentration-time curve up to 24 hours (AUC[0-24 hours]) was calculated from concentration-time data using non-compartmental analysis.
Time Frame: 0 to 24 hours post-dose
Population: Pharmacokinetic analysis set: All randomized patients with evaluable pharmacokinetic data, ie, from which at least one pharmacokinetic parameter could be determined and sampling time information was available, from at least one treatment period.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Groups:
- Indacaterol 150 μg: Patients received Indacaterol 150 μg via the Concept1 dry-powder inhaler only once. There was a washout period of 14-17 days between treatments for patients undergoing pharmacokinetic (PK) assessments; for patients not undergoing PK assessments, the washout period was 7-10 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
Arm/Group | Indacaterol 150 μg | Indacaterol 60 μg | Indacaterol 120 μg
Number analyzed (Participants) | 15 | 14 | 14
pg*hr/mL | 1119.2 (379.1) | 435.8 (245.7) | 849.4 (272.7)

6. Secondary Outcome: Indacaterol Exposure (Cmax) for Each Treatment
Description: All patients fasted for at least 10 hours prior to administration of study medication and continued to fast for at least 4 hours thereafter. Venous blood samples for pharmacokinetic evaluation were collected at 5, 10, 15, and 30 minutes; and 1, 2, 4, 8, and 24 hours post-dose in each treatment period and were analyzed using a LC-MS/MS assay. Maximum (peak) plasma drug concentration after drug administration (Cmax) was calculated from concentration-time data using non-compartmental analysis.
Time Frame: 0 to 24 hours post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Indacaterol 150 μg | Indacaterol 60 μg | Indacaterol 120 μg
Number analyzed (Participants) | 15 | 14 | 14
pg/mL | 150.5 (30.4) | 95.2 (57.3) | 141.7 (55.0)

ADVERSE EVENTS:
Description: Safety population included all randomized patients that received at least one dose of study drug.
Groups:
- Indacaterol 150 μg: Patients received indacaterol 150 μg via the Concept1 dry-powder inhaler (DPI)only once. There was a washout period of 14-17 days between treatments for patients undergoing pharmacokinetic (PK) assessments; for patients not undergoing PK assessments, the washout period was 7-10 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
Arm/Group | Indacaterol 150 μg | Indacaterol 60 μg | Indacaterol 120 μg | Placebo to Indacaterol
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 19/33 | 16/33 | 21/34 | 11/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=33) | Indacaterol 60 μg (N=33) | Indacaterol 120 μg (N=34) | Placebo to Indacaterol (N=35)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 5 | 4 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 15 | 19 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.